CLINICAL TRIAL: NCT06723899
Title: Examining the Effectiveness, and Cost-effectiveness, of CanWork, a Self-management Intervention to Support Women with Breast Cancer to Return to Work
Brief Title: Testing the Effectiveness of a Work Rehabilitation Intervention for Women with Breast Cancer
Acronym: CanWork
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: National Cancer Control Programme, Ireland (Unknown); Royal College of Surgeons, Ireland (Other); University of Galway (Other)
Responsible Party: Principal Investigator, Deirdre Connolly, Professor in Occupational Therapy, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TRI-CFR 23-06
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Self-Management intervention; Occupational Therapy; Self-Efficacy; Return to work; Symptom management
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a cluster randomised control trial. One group will receive the intervention and the other group will receive standard care
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): The intervention arm will receive an online occupational therapy intervention, CanWork, to increase knowledge and skills of women with breast cancer to manage cancer-related symptoms that interfere with return to work. It consists of five, 90-minute group-based modules and an individual meeting between the occupational therapist facilitator and each participant. Each of the group-based modules consists of two components. The first component focuses on education and peer-led discussion of cancer-related symptom management and supports available to manage difficulties in work. Topics covered each week include managing fatigue in work, understanding cancer-related cognitive impairments, strategies for managing physical and mental health in work and effective communication with employers and colleagues.
  Interventions: Other: CanWork
- Comparator group (No Intervention): This group will act as a comparison group to the intervention arm. Study participants (women with breast cancer) in this group will not receive the CanWork intervention but will receive standard supportive care provided in their local community cancer support centre

INTERVENTIONS:
Other: CanWork — CanWork is an online, occupational therapy intervention to develop knowledge and skills to manage cancer-related symptoms that interfere with return to work. It consists of five, 90-minute group-based modules and an individual meeting between the occupational therapist facilitator and each participant. Each of the five-week group-based modules consists of two components: (i) education and peer-led discussion of cancer-related symptom management and supports available to manage difficulties in work and (ii) goal setting to facilitate application of knowledge and skills to work-related activities. Weekly topics include managing fatigue in work, understanding cancer-related cognitive impairments, strategies for managing physical and mental health in work and effective communication with employers and colleagues. The individual meeting between each participant and the occupational therapist is focused on designing a tailored return to work plan for each participant.
  Arms: Intervention arm

SUMMARY:
Women with breast cancer make up a significant proportion of cancer survivors, with more than 43,750 women living with breast cancer in Ireland. However, many women report physical and psychological health difficulties that interfere with their ability to return to work. In Ireland, and internationally, these difficulties are being increasingly recognised, with recent research identifying gaps in rehabilitation services to prepare women with breast cancer to return to work. Collaborating with women with breast cancer, and those who provide health and supportive services to individuals living with cancer in Ireland, an online self-management intervention, CanWork, was developed. CanWork aims to support women with breast cancer to manage the process of returning to work and learn strategies to manage post-treatment health-related difficulties. CanWork also provides information on workplace entitlements. This intervention was trialled with women with breast cancer in 2021, who reported that the programme gave them confidence to return to work and that the content was relevant. This study will include a larger group of women with breast cancer to determine if CanWork is effective in supporting return to work. To do this, 248 women with breast cancer will be included in the study, half of whom will receive CanWork and the results will be compared with women who do not receive the intervention. Having a programme that is financially viable is important and therefore the costs involved in running and attending the intervention will also be calculated. Should this study demonstrate that CanWork is effective in supporting women with breast cancer to return to work, the study team will collaborate with cancer services in Ireland to make the programme available nationally.

DETAILED DESCRIPTION:
The importance of supporting return to work (RTW) following a cancer diagnosis is increasingly recognised nationally and internationally. Other countries including the United Kingdom, Canada, and the United States, have also identified the importance of addressing work outcomes for those living with and beyond cancer. The goal for many cancer survivors is to optimise quality of life, including return to work. A recent report by the European Commission recommended that assessment and interventions for enhancing return to work for those with cancer should be integral parts of the survivorship pathway. As survivor numbers continue to increase the economic benefit of individuals returning to work will be considerable.

Breast cancer is now the most common cancer worldwide. In Ireland, the National Cancer Strategy (2017-2026) identified that 23% of all cancer survivors are comprised of women with breast cancer. The impact of disease and treatment-related side effects on work ability of women with breast cancer include cancer-related fatigue, pain, reduced cognitive function, anxiety, and depression. Therefore research is recommended for the development and evaluation of interventions to support women living with and beyond breast cancer to return to, and manage cancer related symptoms at, work.

CanWork is an online, occupational therapy self-management intervention that was designed in collaboration with women with breast cancer, healthcare professionals, cancer service providers and Health Service Executive staff with responsibility for development and delivery of cancer services in Ireland. Self-efficacy is the underlying theory of self-management interventions. Self-efficacy is the belief individuals have in their ability to change and take the necessary actions to make those changes. Perceived self-efficacy forms the basis of any decision to act and is defined as the perception of one's own ability to implement behaviours to attain designated types of outcomes such as improved health and well-being.

The primary aim of CanWork is to facilitate development of knowledge and skills to manage cancer-related symptoms that interfere with return to work. It consists of five, 90-minute group-based meetings and a once-off single individual meeting between the occupational therapist facilitator and each participant. Each of the group-based sessions consists of two components. The first component focuses on education and peer-led discussion of cancer-related symptom management and supports available to manage difficulties in work. The topics covered each week include managing fatigue in work, understanding cancer-related cognitive impairments, strategies for managing physical and mental health in work and effective communication with employers and colleagues.

Feasibility testing of CanWork demonstrated strong uptake for, and acceptability of, the intervention. The aim of this study, therefore, is to test the effectiveness of the CanWork intervention in facilitating women with breast cancer to return to work.

Methods

Study design A Cluster randomised trial (CRT) will be used to test the effectiveness of the CanWork intervention. The CRT will be carried out within the Medical Research Council (MRC) Framework for the development and evaluation of complex interventions to improve health outcomes for individuals with chronic health difficulties. The CONSORT guidelines extension for cluster randomised trials for the design and reporting of randomized controlled trials at all stages from recruitment of cancer centres (study clusters) and individual participants, randomisation, data collection, analysis and reporting will be used. (www.equator-network.org)

The units of randomisation for this study are Community Cancer Support Centres. In Ireland Community Cancer Support Centres (CCSC) are recognised as an essential part of provision of support for individuals with cancer, their families and carers. They provide a range of services from the provision of information, psychological support and survivorship programmes, to complementary therapies, yoga, relaxation classes, support groups, financial advice and drop-in services. CCSC operate in the charity sector and mainly rely on fund-raising activities to fund delivery of their services but they also receive project-based governmental funding.

Study sample The sample size required for this study is 248 women with breast cancer. This is based on detecting a 22% difference in return-to-work rates between the control and intervention clusters.

Data collection

This study will use two primary outcome measures:

Return to work: Yes/No. Return to Work Self-efficacy (RTW-SE) questionnaire

Secondary measures will examine readiness to return to work, self-efficacy for managing cancer-related symptoms that interfere with work, breast cancer specific quality of life measures, and a log book of work attendance. Cost effectiveness measures include EQ-5D-5L, ICECAP-A capability measure, work log book and cost of intervention delivery.

Data analysis

Quantitative Data Analysis

Analysis will be based primarily on intention-to-treat comparing outcomes at baseline and post-intervention follow-up periods. A per protocol analysis will be conducted as sensitivity analysis only. Descriptive analyses will include frequencies (%), means (standard deviation, 95%CI) and medians (inter-quartile range, IQR) where appropriate. A baseline table of characteristics for all participants recruited and by sites recruiting will be presented to ensure balance achieved with randomisation. Numbers of those recruited from participating CCSC, numbers (percentage) of those randomised and enrolled into intervention, and numbers (percentage) adhering to the intervention and retained in the study will be examined.

Qualitative data analysis All interviews will be audiotaped and transcribed verbatim. Analysis will be carried out using a computer software package, NVivo (available through TCD IS services). A content analysis approach will be used to explore commonalities between participants on their experiences of the intervention and to identify differences in experiences and opinions of the intervention. Within a content-analysis framework, both a deductive and inductive approach will be used for the analysis to identify new findings related to the CanWork intervention (inductive analysis) and to compare the findings of this study to previously reported research on work-focused interventions (i.e. deductive analysis).

Cost effectiveness analysis The health economics analysis will consist of trial-based economic evaluation and will incorporate cost utility analysis to compare the alternative strategies: (1) the CanWork self-management intervention; and (2) usual practice. The economic evaluation will be undertaken in a manner consistent with the guidelines issued by Health Information and Quality Authority (HIQA) for the evaluation of healthcare interventions and technologies in Ireland. The basic tasks of the evaluation are to identify, measure, value and compare the costs and outcomes of the alternatives being considered.

ELIGIBILITY:
Inclusion Criteria:

* Women with confirmed diagnosis of breast cancer
* Women with breast cancer who were in paid employment prior to their cancer diagnosis
* Women with breast cancer who have completed adjuvant oncology treatment (excluding hormone therapy, targeted and biological therapies) within the last 12 months
* Women with breast cancer who have capacity to participate in a six-week online occupational therapy intervention

Exclusion Criteria:

* Women with metastatic breast cancer
* Women with breast cancer who were not in paid employment prior to their cancer diagnosis
* Women with breast cancer who have decided not to return to work following completion of cancer treatment
* Women with breast cancer who have co-morbidity that would interfere with capacity to participate in a six-week online occupational therapy intervention

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Return to work: Yes/No. | From enrolment to 12-months following enrolment
  The primary outcomes measure used in the feasibility study of CanWork was a self-report binary question of "Return to Work (RTW): Yes/No. This measure was identified in a systematic review as the most commonly used work-related measure in the included studies. RTW refers to any work resumption irrespective of number of hours a participant worked before their diagnosis. Participants will be asked immediately post-intervention, at three, six and 12-month follow-up periods if they have returned to work, on what date they returned and number of hours/week currently working
Return to Work Self-efficacy (RTW-SE) questionnaire | From enrolment to 12-months following enrolment
  The RTW-SE measure is a short ten-item questionnaire that asks participants to rate their level of confidence on a Likert scale of 1-10 to manage physical, psychological and emotional demands of work. Recent research has found that both the baseline RTW-SE score and subsequent increases in the RTW-SE score during return-to-work interventions are robust predictors of return to work.

SECONDARY OUTCOMES:
Readiness to return to work | From enrolment to 12-months following enrolment
  Participants will rate their current perceived readiness to return to work on a 10-point Likert scale: 0 (not at all ready) to 10 (extremely ready).
Return to Work log book | From enrolment to 12-months following enrolment
  All participants (intervention and control group) who have returned to work will be required to keep a work-related logbook over a 12-month period following enrolment into the CanWork study. This logbook will record any absences (planned or unplanned) from work for cancer-related reasons. The following information will be collected:
  Dates of absenteeism Reason for absenteeism Date returned to work Total time absent from work
EORTC QLQ-30 | From enrolment to 12-months following enrolment
  Health related quality of life will be measured using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) with the relevant subscale for breast cancer QLQ-BR23. The EORTC-QLQ-C30 includes 30 items embedded over nine scales: five functional scales (physical, role, cognitive, emotional, and social functioning), three symptom scales (fatigue, pain, nausea and vomiting), and a global health status quality of life scale. Six single-items assess financial difficulties and symptoms commonly reported by those living with and beyond cancer: dyspnoea, insomnia, appetite loss, constipation and diarrhoea. The QLQ-BR23 questionnaire comprises of 23-items and is categorised into functional scales and symptom scales. Functional scales include items on body image, sexual functioning, sexual enjoyment, and future perspective. Future perspective explores the extent to which a participant is worried about their health in the future.
PROMIS Self-Efficacy for Managing Symptoms | From enrolment to 12-months following enrolment
  The PROMIS Self-Efficacy for Managing Symptoms is an eight-item measure that examines participants' confidence in managing their symptoms in different settings (home, work and public places) and in preventing their symptoms from interfering with their personal activities, work and relationships. This measure has been calibrated across a number of different chronic diseases and demonstrates strong internal consistency and validity.

OTHER OUTCOMES:
ICECAP-A (ICEpop CAPability measure for Adults) | From study enrolment to 12-months following enrolment
  ICECAP-A is designed to assess overall quality of life and well-being of adults. It focuses on broader life aspects rather than just health-related factors. The measure is based on the concept of capability, which considers what individuals are able to do in their lives, encompassing a range of attributes that contribute to a fulfilling life. ICECAP-A evaluates five key dimensions of capability: Stability Attachment, Autonomy, Achievement and Enjoyment. Respondents rate their level of capability in each dimension, providing a comprehensive picture of their overall well-being. The ICECAP-A total score will be converted to a utility score to assess cost effectiveness of CanWork.

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Connolly, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (2):
- Ireland (2):
  - Cancer Care West, Galway
  - Solas Cancer Support Centre, Waterford

IPD SHARING:
Plan to Share IPD: No
Ethical approval has not been obtained to share IPD

REFERENCES:
- [Derived] Pallin ND, Algeo N, O'Connor ME, Connolly H, Lowry M, Bennett K, Gillespie P, Hobbins A, Gallagher P, Mullen L, Lyons KD, McHugh SM, Connolly D. A cluster randomised controlled trial to test the effectiveness and cost-effectiveness of a self-management intervention to support women with breast cancer to return to work: A study protocol. Contemp Clin Trials. 2025 Dec 15;161:108185. doi: 10.1016/j.cct.2025.108185. Online ahead of print. PMID 41407101